CLINICAL TRIAL: NCT06392230
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY IN HEALTHY ADULT MALE PARTICIPANTS TO ASSESS THE MASS BALANCE, ABSOLUTE BIOAVAILABILITY, FRACTION ABSORBED, AND PHARMACOKINETICS OF [14C]PF-06821497 USING A 14C-MICROTRACER APPROACH
Brief Title: A Study to Learn How the Medicine Called [14C] PF-06821497 is Taken up Into and Removed From the Body.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C2321007; 2023-508371-36-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-04-12; First posted 2024-04-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
Keywords: Absorption; Distribution; Metabolism; Elimination; ADME (Absorption, Distribution, Metabolism, and Excretion); Pharmacokinetics; Bioavailability; Fraction absorbed; Mass balance; Healthy Males; Enhancer of zeste homolog 2 (EZH2) inhibitor
MeSH Terms: interventions — PF06821497

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort 1 (Experimental): Participants will receive one dose of [14C] PF-06821497 by mouth in Period 1. After a washout, participants will receive one dose of PF-06821497 by mouth and one intravenous (IV) infusion of [14C] PF-06821497 in Period 2
  Interventions: Drug: Oral [14C] PF-06821497; Drug: Oral PF-06821497; Drug: IV [14C] PF-06821497

INTERVENTIONS:
Drug: Oral [14C] PF-06821497 — A single oral dose of [14C] PF-06821497 will be administered as an extemporaneous suspension in Period 1
Drug: Oral PF-06821497 — A single oral dose of PF-06821497 will be administered as an extemporaneous oral suspension in Period 2
Drug: IV [14C] PF-06821497 — A single IV infusion of [14C] PF-06821497 will be administered at the Tmax after administration of the unlabeled oral dose of PF-06821497 in Period 2

SUMMARY:
The purpose of this study is to learn how a certain amount of [14C] PF-06821497 is taken up into the bloodstream and removed from the body.

The study is seeking participants who are:

* Males aged 18 years or older.
* Are confirmed to be healthy after performing some medical and physical tests.
* Weigh more than 50 kilograms and have a body mass index of 16 to 32 kg per meter squared.

The study consists of two parts. In part one, all participants will receive one full dose of [14C]PF-06821497 by mouth. Part two will begin at least 14 days after the dose in part one. In part two participants will receive one full dose of PF-06821497 by mouth and one small dose of [14C]PF-06821497 by intravenous (IV) infusion. IV infusion will be directly injected into the veins.

To understand how the medicine is processed in the body, samples of blood, urine, and feces will be collected after each dose is given. This will help understand:

* How much PF-06821497 is taken up into the bloodstream when taken by mouth compared to the dose given by IV
* How the body removes it from the bloodstream.

Participants will take part in the study for about 11 weeks, including the initial evaluation and follow-up periods.

ELIGIBILITY:
Key eligibility criteria for this study include, but are not limited to the following:

Inclusion Criteria:

* Male participants aged 18 years at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body mass index (BMI) of 16-32 kg/m2; and a total body weight of >50kg (110lb)
* Participants who are willing to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, prior bariatric surgery, ileal resection, inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease).
* Chronic liver diseases including alcoholic liver disease, viral hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency, human immunodeficiency virus, or other chronic liver disease.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* Total [14C] radioactivity measured in plasma at screening exceeding 11 mBq/mL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactivity in urine, feces, and total excreta (urine + feces) as percentage of total radioactive dose administered | Period 1 pre-dose to maximum Day 14
  To characterize the extent of excretion of total radioactivity in urine and feces following administration of a single oral dose of [14C]PF-06821497
Metabolic profiling/identification and determination of relative abundance of [14C]PF-06821497 and the metabolites of [14C]PF-06821497 in plasma, urine, and feces | Period 1 pre-dose to maximum Day 14
  Amount of metabolites of [14C]PF-06821497 in plasma, urine, and feces

SECONDARY OUTCOMES:
Absolute oral bioavailability (F) of [14C]PF-06821497 | Period 2 pre-dose to maximum Day 5
  To determine the absolute oral bioavailability (F) of PF-06821497 by comparing AUCinf following administration of a single oral dose of PF-06821497 to a single IV microtracer of [14C]PF 06821497
Fraction of [14C]PF 06821497 dose absorbed (Fa) | Period 1 pre-dose to maximum Day 14; Period 2 pre-IV dose to maximum Day 5
  To determine the fraction of the dose absorbed (Fa) following administration of a single oral dose of [14C]PF 06821497 from total urinary radioactivity of [14C]PF 06821497 in Period 1 and IV microtracer microdose administration of [14C]PF 06821497 in Period 2
AUClast of total radioactivity and PF-06821497 in plasma | Period 1 pre-dose to maximum Day 14
  To quantify plasma area under the concentration versus time curve (AUClast) of PF-06821497 and total radioactivity following administration of a single oral dose of [14C]PF-06821497.
Cmax of total radioactivity and PF-06821497 in plasma | Period 1 pre-dose to maximum Day 14
  To quantify plasma peak concentration (Cmax) of PF-06821497 and total radioactivity following administration of a single oral dose of [14C]PF-06821497.
Tmax of total radioactivity and PF-06821497 in plasma | Period 1 pre-dose to maximum Day 14
  To quantify plasma time of peak concentration (Tmax) of PF-06821497 and total radioactivity following administration of a single oral dose of [14C]PF-06821497.
AUCinf of total radioactivity and PF-06821497 in plasma | Period 1 pre-dose to maximum Day 14
  If data permits, to quantify plasma area under the concentration versus time curve extrapolated to infinity (AUCinf) of PF-06821497 and total radioactivity following administration of a single oral dose of [14C]PF-06821497.
t½ of total radioactivity and PF-06821497 in plasma | Period 1 pre-dose to maximum Day 14
  If data permits, to quantify plasma half-life (t½) of PF-06821497 and total radioactivity following administration of a single oral dose of [14C]PF-06821497.
AUClast of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  To quantify plasma area under the concentration versus time curve (AUClast) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
Cmax of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  To quantify plasma peak concentration (Cmax) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
Tmax of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  To quantify plasma time of peak concentration (Tmax) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
t½ of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  If data permits, to quantify plasma half-life (t½) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
AUCinf of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  If data permits, to quantify plasma area under the concentration versus time curve extrapolated to infinity (AUCinf) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
CL of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  If data permits, to quantify plasma clearance (CL) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
Vss of [14C]PF-06821497 in plasma | Period 2 pre-dose to maximum Day 5
  If data permits, to quantify plasma volume of distribution at steady-state (Vss) of PF-06821497 following administration of a single, IV, microtracer of [14C]PF-06821497.
Number of participants with treatment emergent clinically significant laboratory abnormalities | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal ECG measurements | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal vital measurements | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment emergent clinically significant abnormal physical examination | Both cohorts from pre-dose to 28 days post-dose
Number of participants with treatment-emergent adverse events (AEs) or serious adverse events (SAEs) | Both cohorts from pre-dose to 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321007